CLINICAL TRIAL: NCT00001626
Title: A Randomized Trial of Antithymocyte Globulin and Cyclosporine Versus Cyclophosphamide and Cyclosporine in the Treatment of Severe Aplastic Anemia
Brief Title: Comparing Therapies for the Treatment of Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 970117; 97-H-0117
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Severe Aplastic Anemia; Immunosuppression
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): D1-4 cyclophosphamide 50 mg/kg IV, then cyclosporine starting on d14 at 12 mg/kg/d for 6 months
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine
- B (Experimental): ATG at 40 mg/kg/d for 4 days then cyclosporine at 12 mg /kg/d for 6 months
  Interventions: Drug: antithymocyte globulin; Drug: cyclosporine

INTERVENTIONS:
Drug: antithymocyte globulin — antithymocyte globulin
  Arms: B
Drug: cyclophosphamide — cyclophosphamide
  Arms: A
Drug: cyclosporine — cyclosporine

SUMMARY:
Severe Aplastic Anemia (SAA) is a rare and very serious blood disorder in which the bone marrow stops producing the cells which make up blood; red blood cells, white blood cells, and platelets.

Researchers believe this is caused by an autoimmune reaction, a condition in which the natural defense system of the body begins attacking itself. In SAA the immune system begins attacking the bone marrow. Red blood cells are responsible for carrying oxygen to all of the organ systems in the body, and low numbers (anemia) can cause difficulty breathing and fatigue. Platelets are responsible for normal blood clotting and low numbers can result in easy bruising and bleeding which can be deadly. White blood cells are responsible for fighting infections, and low numbers of these can lead to frequent infections, the most common cause of death in patients with aplastic anemia.

SAA can be treated by bone marrow transplant (BMT) or by drugs designed to slow down the immune system (immunosuppressants). BMT can be successful, but it requires a donor with matched bone marrow, making this therapy available only to a few patients. BMT with unmatched bone marrow can fail and cause dangerous side effects.

Presently, the two drugs used to treat SAA by slowing down the immune system (immunosuppression) are antithymocyte globulin (ATG) and cyclosporin A (CSA). When used in combination these two drugs can improve most patients condition. However, one third of the patients who respond to this therapy experience a relapse of SAA. In addition, some patients treated with ATG/CSA can later develop other disorders of the blood.

Recently, researchers have found that another immunosuppressive drug called cyclophosphamide, has been successful at treating patients with SAA. In addition, patients treated with cyclophosphamide do not experience relapses or develop other disorders of the blood.

In this study researchers would like to compare the combinations of antithymocyte globulin (ATG) and cyclosporin A (CSA) to cyclophosphamide and cyclosporin A (CSA) for the treatment of SAA.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a disorder with a poor prognosis if untreated. Current accepted therapeutic strategies include bone marrow transplantation (BMT) and immunosuppression, both offering cure or amelioration in the majority of patients. Although BMT is successful using human leukocyte antigen (HLA) matched sibling bone marrow, the 25% probability of finding an HLA identical sibling within a family renders this approach available to only a minority of patients. BMT utilizing HLA-matched, unrelated donors carries a high risk of treatment failure along with considerable toxicity. While combined immunosuppression with both antithymocyte globulin (ATG) and cyclosporine A (CSA) produces hematologic improvement in most patients, relapse is common, occurring in about a third of responders. Late evolution of aplastic anemia to other serious hematologic disorders is a significant problem following successful treatment with ATG/CSA with paroxysmal nocturnal hemoglobinuria (PNH) occurs in approximately 13%, myelodysplasia in about 10%, and acute leukemia in about 7%. Recently, results of immunosuppression in SAA with another potent immunosuppressive agent, cyclophosphamide, were reported in 10 patients. In this small group, the overall response rate was similar to that seen with ATG/CSA, but relapse and late clonal disease were not seen during a median follow-up of greater than 10 years. In the larger randomized trial proposed here, we will compare sustained hematologic response rates to either conventional immunosuppression with ATG/CSA or high dose cyclophosphamide and CSA. Secondary endpoints include response duration, event free survival, and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

Severe aplastic anemia confirmed at NIH by:

1. Bone marrow cellularity less than thirty percent (excluding lymphocytes).
2. At least two of the following:

Absolute neutrophil count less that 500/mm(3);

Platelet count less than 20,000/mm(3);

Reticulocyte count less than 60,000/mm(3).

EXCLUSION CRITERIA:

Serum creatinine greater than to 2.5 mg/dl.

Cardiac ejection fraction less than 45% by MUGA.

Underlying carcinoma (except local cervical, basal cell, squamous cell or melanoma).

Current pregnancy or unwilling to take oral contraceptives.

Diagnosis of Fanconi anemia or other congenital bone marrow failure syndromes.

Evidence of a clonal disorder on cytogenetics.

HIV positivity.

Inability to understand the investigational nature of the study.

Patients who are moribund or have hepatic, renal, cardiac, metabolic or other concurrent diseases of such severity that death within 7-10 days is likely.

Previous treatment with ATG, or cyclophosphamide.

Ages: 15 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1997-06-02 (Actual); Primary Completion 2001-02-20 (Actual); Study Completion 2008-03-03 (Actual)

PRIMARY OUTCOMES:
Compare the sustained response proportions among patients with SAA treated with immunosuppressive therapy with either ATG/CSA or high dose cyclophosphamide and CSA. | 12 weeks.

SECONDARY OUTCOMES:
Overall and event-free survival. | 12 months
Response duration. Evolution to PNH, myelodysplasia, and active leukemia. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-H-0117.html